CLINICAL TRIAL: NCT02627651
Title: The Cardiac Autonomic System Response to Activity and Cognitive Tasks in Children Post Acquired Brain
Brief Title: The Cardiac Autonomic System Response to Activity and Cognitive Tasksinjury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Alyn
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

ARMS (2):
- brain injury (Experimental): children post brain injury
  Interventions: Other: cognitive and motor assignments
- controls (Active Comparator): children typically developed age matched
  Interventions: Other: cognitive and motor assignments

INTERVENTIONS:
Other: cognitive and motor assignments — walking on treadmill, performing cognitive assignment; and performing the cognitive assignment while walking .

SUMMARY:
18 children post acquired brain injury and 18 typically developed controls matched for age and gender.

All children aged 10-18 yrs who understand simple commands.

Tools:

1. Heart rate monitor
2. Six minute walk test
3. The behavior rating inventory

Method:

1. At the introductory visit the child will be asked to walk for six minutes, to sit and perform a cognitive test and then to walk on a treadmill for 5 seconds.
2. At the second visit the child will be asked to go on the treadmill for 5 minutes and at the same time to perform the cognitive assignment; After a rest the child will be asked to walk on the treadmill for 5 minutes and at the end to perform the cognitive assignment .

ELIGIBILITY:
Inclusion Criteria:

aged 10-18 understand simple commands walk independently

Exclusion Criteria:

Canot understand simple commands

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Heart rate | 5 min
Heart rate variability- time domain measures | 5 min
Heart rate variability- frequency domain measures | 5 min

CONTACTS AND LOCATIONS:
Locations (1):
- Alyn Pediatric and Adolesencent Rehabilitation Center, Jerusalem, Israel